CLINICAL TRIAL: NCT00832286
Title: Longitudinal Study of the Human Intestinal Microbiome Before and After Antibiotic Administration
Brief Title: Longitudinal Study of the Human Intestinal Microbiome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 07-0053
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2011-02-08

CONDITIONS: Dysbacteriosis
Keywords: genomic techniques; intestinal microbiome
MeSH Terms: conditions — Dysbiosis | interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cipro (Experimental): At Week 12, subjects will receive a 3-day course of oral Ciprofloxacin 500 mg every 12h.
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: Ciprofloxacin — Licensed medication, dose: 500 mg every 12 hours for 3 days.

SUMMARY:
The purpose of this study is to identify the human intestinal microbiota (microbes that live inside and on human bodies) in healthy adults over a 6-month period and to study the effect of an antibiotic on the intestinal microbiota. Participants will include up to 60 healthy adult subjects, ages 18-45 years, from the Baltimore and University of Maryland communities. Study procedures will include providing multiple stool samples throughout the study. Participants will take a licensed antibiotic, Ciprofloxacin, for 3 days. Participants may be involved in study related procedures for up to 7 months.

DETAILED DESCRIPTION:
The purpose of this study is to describe the intestinal microbiomes of a cohort of healthy adult subjects over a 6-month period of time. Many questions about the human microbiota exist. Previous studies have shown that the differences among individuals are greater than the differences among different sampling sites in a single individual. Up to 60 healthy adult subjects, ages 18-45 years, from the Baltimore and University of Maryland Baltimore communities will be recruited and screened to document their health status. A brief medical history, including recent travel and antibiotic use, will be recorded. Subjects will provide a stool specimen for genomic analysis of the intestinal microbiome over a 6-month period at the following intervals: Day 0, Week 1, Week 2, Week 3, Week 4, Week 8, Week 12, Week 13, Week 14, Week 15, Week 16, Week 20, and Week 24. At Week 12, subjects will receive a 3-day course of oral Ciprofloxacin 500 mg every12 hours. Weekly stool specimens will be obtained beginning with the first day of antibiotic use and for 4 Weeks thereafter. Then monthly specimens of stool and other sites will be resumed at Week 16. The primary objective is to define the human intestinal microbiome in healthy adults in a longitudinal fashion. The secondary objective is to define the re-colonization of the intestine after treatment with a broad-spectrum antibiotic using comprehensive genomic techniques. Each subject will participate in the study for up to 7 months.

ELIGIBILITY:
Inclusion Criteria:

-Male or female, ages 18 to 45 years, inclusive. -Healthy as determined by screening medical history, medication history, and absence of acute illness such as gastrointestinal or respiratory infection. -Capable of understanding, consenting and complying with the entire study protocol. -Provide voluntary written Informed Consent. -Females of childbearing potential are required to utilize an appropriate method of contraception [abstinence, oral contraceptives, IUD, condoms with spermicidal foam, surgical sterilization depots and injectable contraceptives, or diaphragms with spermicidal jelly or cream] 30 days prior to the Week 12 visit.

Exclusion Criteria:

-Chronic diarrhea, inflammatory bowel disease, irritable bowel syndrome, or other gastrointestinal disorder, gastrointestinal surgery (except appendectomy, polypectomy, or herniorraphy), or severe chronic illness such as major organ failure, diabetes, HIV/AIDS. -Female who is pregnant or lactating; or a female subject with a positive urine pregnancy test determined at the Week 12 visit. -History of hypersensitivity to Ciprofloxacin, any member of the quinolone class of antimicrobial agents, or any compound of the product. -History of tendinitis or tendon rupture. -History of seizures other than febrile seizure as a young child. -Treatment with antibiotics within one month before the initial specimen collection. -History of clinically significant acute or chronic illness or other condition requiring chronic medication therapy (including systemic but not intranasal steroids), except for birth control pills, inhalers, anti-anxiety or anti-depression medications. -History of cardiac rhythm abnormalities or QT prolongation or a family history of cardiac rhythm abnormalities or sudden unexplained death. -History of current or past use of theophylline for asthma or tizanidine, due to known interaction with Ciprofloxacin. -History of spasticity (due to the potential for requiring tizanidine treatment), asthma, chronic bronchitis, emphysema, and other lung diseases (due to potential for requiring theophylline [or dimethylxanthine] treatment). -Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-07-23 (Actual); Primary Completion 2010-09-24 (Actual); Study Completion 2011-01-11 (Actual)

PRIMARY OUTCOMES:
Analysis of GI microbial community composition using the Affymetrix PhyloChip Platform. | Analysis.
Isolation of Genomic DNA from stool samples. | Weekly stool samples will be obtained for over a 6-month period at the following intervals: Day 0, Weeks 1, 2, 3, 4, 8, 12, 13, 14, 15, 16, 20, and 24.
Surveys of GI microbiome diversity using 16S rDNA analysis at the Institute of Genome Sciences. | Analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland, United States